CLINICAL TRIAL: NCT03553810
Title: Role of ARNi in Ventricular Remodeling in Hypertensive LVH
Acronym: REVERSE-LVH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart Centre Singapore (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018/2182
Record Dates: First submitted 2018-04-04; First posted 2018-06-12 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Hypertensive Heart Disease
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination; Valsartan

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Entresto (valsartan/sacubitril) 100mg once a day
  Interventions: Drug: Entresto
- Controlled Arm (Active Comparator): Valsartan 40mg once a day
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Entresto — Entresto (Valsartan/sacubitril) 100mg once a day, up-titrating to 200mg or maximum 400mg to achieve target systolic blood pressure below 140 mmHg, over a duration of 52 weeks. If necessary, amlodipine and/or hydrochlorothiazide may be added to achieve target systolic blood pressure.
  Other Names: Valsartan/sacubitril
  Arms: Treatment Arm
Drug: Valsartan — Valsartan 40mg once a day, up-titrating to 80 or maximum 160 mg to achieve target systolic blood pressure below 140mmHg, over a duration of 52 weeks. If necessary, amlodipine and/or hydrochlorothiazide may be added to achieve target systolic blood pressure.
  Arms: Controlled Arm

SUMMARY:
In Singapore, hypertension is very common in the adult population. Hypertensive heart disease is a leading cause of heart failure and cardiovascular death. Current management relies primarily on achieving blood pressure targets. However, the optimal blood pressure goals are controversial and there are inherent difficulties in measuring blood pressure using external devices applied to peripheral arteries. As a result of (usually longstanding) hypertension, the heart thickens (i.e. hypertrophies) to maintain function. Ultimately, HF may occur due to long standing energy deficits, muscle injury/death and diffuse interstitial fibrosis (heart muscle scarring). In an ongoing study (REMODEL, ClinicalTrial.gov Identifier NCT02670031), we have been able to undertake preliminary analyses with respect to factors associated with the development of fibrosis. In this randomize controlled trial, we will be examining a novel therapy that has the potential to induce regression cardiac hypertrophy and fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Increased left ventricular mass on cardiovascular magnetic resonance (based on established local age- and sex-specific CMR ranges)
* Essential hypertension

Exclusion Criteria:

* Known secondary causes of hypertension
* Previous intolerance to angiotensin receptor blockers
* History of heart failure
* Stage IV/V chronic renal disease (eGFR < 30ml/min/1.73m2)
* Patients with serum potassium > 5.2 mmol/L (mEg/L) at Visit 1
* History of cardiovascular events (myocardial infarction, strokes and transient ischemic attacks)
* Known atrial fibrillation
* Being unable to understand or comply with study procedures (including CMR)
* History or presence of any other disease with a life expectancy of < 3 years
* Pregnant or nursing (lactating) women

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Fibrosis volume | 52 weeks
  A difference in terms of change in interstitial volume from baseline following 52 weeks of treatment. Extracellular volume fraction (ECV) will be quantified from native and post-contrast myocardial T1. Fibrosis volume is defined as ECV x myocardial volume and indexed to body surface area (ml/m2)

SECONDARY OUTCOMES:
Left ventricular mass measured on CMR | 52 weeks
  Changes from baseline in left ventricular mass, indexed to body surface area (g/m2).
Biomarker/biochemistry | 52 weeks
  Identify potential markers as indicators of cardiac structural effects of ARNi and ARB

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee V, Zheng Q, Toh DF, Pua CJ, Bryant JA, Lee CH, Cook SA, Butler J, Diez J, Richards AM, Le TT, Chin CWL. Sacubitril/valsartan versus valsartan in regressing myocardial fibrosis in hypertension: a prospective, randomized, open-label, blinded endpoint clinical trial protocol. Front Cardiovasc Med. 2023 Aug 22;10:1248468. doi: 10.3389/fcvm.2023.1248468. eCollection 2023. PMID 37674806